CLINICAL TRIAL: NCT02229682
Title: Mild-dose Intensity-modulated Radiation Treatment for Stage IE/IIE Extranodal Nasal-type NK/T-cell Lymphoma With Complete Remission Tumor After Combination of Gemcitabine, Oxaliplatin, and Asparaginase (GELOX) Chemotherapy:a Phase II Study
Brief Title: Mild-dose IMRT for Early-staged Extranodal Nasal-type NK/T-cell Lymphoma With CR Tumor After GELOX Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yujing ZHANG, MD/PhD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-NKTRT-01
Record Dates: First submitted 2014-08-27; First posted 2014-09-01 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma,; Non-Hodgkin Lymphoma,; Extranodal NK/T-cell Lymphoma,Nasal-type,
Keywords: extranodal NK/T-cell lymphoma,nasal-type,; radiotherapy,; intensity-modulated radiation treatment,; asparaginase-based chemotherapy,; loco-regional control,; survival
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mild-dose IMRT (Experimental): Experimental: Mild-dose of 46Gy with IMRT
  Drug:
  gemcitabine：1250mg/m2 (iv drip) on days 1, oxaliplatin: 85 mg/m2 (iv drip) on day 1, and pegaspargase: 2500 IU/m2 (intramuscular injection) on day 1. Cycle is repeated every 14 days
  IMRT： IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 46.2 grays (Gy) in 22 fractions.
  Interventions: Radiation: Mild-dose IMRT

INTERVENTIONS:
Radiation: Mild-dose IMRT — IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 46.2 grays (Gy) in 22 fractions.
  Other Names: Mild-dose intensity-modulated radiation treatment

SUMMARY:
This study is to make sure whether reduced-dose radiation treatment is sufficient to control the disease in patients with early-staged extranodal nasal-type NK/T-cell lymphoma, who have got complete remission tumor after chemotherapy in a new and more effective asparaginase-based GELOX regimen

DETAILED DESCRIPTION:
Definitive radiotherapy(RT) is mainstay in combined-modality treatment for patients with early-staged extranodal nasal-type NK/T-cell lymphoma(ENKTL),it can be used upfront or after short courses of chemotherapy. The typical dose of RT is recommended as 50-56Gy in conventional fractionations with 3 dimensional conformal RT or intensity-modulated radiation treatment(IMRT). Asparaginase-based chemotherapy regimens are being investigated, and primary results showed superior to previous anthracycline-based (eg. CHOP) chemotherapy. GELOX is a new asparaginase-based chemotherapy regimen designed and published in our institute, and the rate of complete remission(CR) is well improved. We hypothesis the reduced-dose radiation treatment(IMRT in 46Gy) is sufficient to control the disease in patients with early-staged ENKTL, who have got CR after GELOX chemotherapy, and to validate in this phase II study.

1. Patients:

   * All patients should sign a written informed consent form before enrollment, and the study should be approved by the Sun Yat-sen University Cancer Center Ethics Board.
   * Baseline of patients: Computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, and bilateral bone marrow aspiration or biopsy. Positron emission tomography-CT scans (optional). Epstein-Barr virus (EBV) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA).
   * Recheck before and after GELOX chemotherapy and IMRT: Epstein-Barr virus (EBV) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA), computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, positron emission tomography-CT scans (optional).
2. Treatment Protocol:

   1. The GELOX regimen consist of the following drugs: gemcitabine：1250 mg/ m2 on days 1,iv drip; oxaliplatin：85 mg/m2 on day 1, iv drip; pegaspargase: 2500 IU/m 2 daily on day 1,intramuscular. The treatment cycle is repeated every 14 days.
   2. IMRT is delivered using 6-8MeV linear accelerator using extended involved-field intensity-modulated radiation treatment planning. The RT dose is 46.2 grays (Gy) in 22 fractions, and a simultaneous-boost method is used.

      * We assign gross tumor volume (GTV) to 46.2Gy/22F, which is delineated according to the initial gross tumor volume identified with imaging and physical examination, including the primary tumor and involved regional lymph nodes.
      * The high-risk clinical target volume (CTV1) is assigned to 41.8Gy/22F, which is delineated including the first batch of adjacent structures around GTV, and lymph node group apt for involvement according to clinical feature of individual tumors.
      * The low-risk clinical target volume (CTV2) is assigned to 36.3Gy/22F, which is delineated including the extrapolated structures outside of CTV1 sites, and LN groups adjacent to CTV1 LN groups.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-75years
* Ann Arbor stage IE,or stage IIE with cervical lymph node involvement
* at lease one measurable lesion
* received GELOX chemotherapy and got CR before radiotherapy
* Eastern CooperativeOncology Group performance status of 0 to 2
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria,
* got non-CR after GELOX chemotherapy before IMRT,
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol,
* primary lesion not from the upper aerodigestive tract

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
loco-regional tumor control | every 3 months after IMRT for 2 years, and then every 6 months for the next 3 years.
  loco-regional tumor control was examined with physical examination and image methods.

SECONDARY OUTCOMES:
progression-free survival(PFS) | every 3 months after IMRT for 2 years, and then every 6 months for the next 3 years
  progression-free survival(PFS): time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first
overall survival(OS) | every 3 months after IMRT for 2 years, and then every 6 months for the next 3 years
  overall survival (OS): time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Yujing Zhang, MD/PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Dept. Radiation Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wang L, Wang ZH, Chen XQ, Li YJ, Wang KF, Xia YF, Xia ZJ. First-line combination of gemcitabine, oxaliplatin, and L-asparaginase (GELOX) followed by involved-field radiation therapy for patients with stage IE/IIE extranodal natural killer/T-cell lymphoma. Cancer. 2013 Jan 15;119(2):348-55. doi: 10.1002/cncr.27752. Epub 2012 Jul 18. PMID 22811078
- [Background] Gregoire V, Ang K, Budach W, Grau C, Hamoir M, Langendijk JA, Lee A, Le QT, Maingon P, Nutting C, O'Sullivan B, Porceddu SV, Lengele B. Delineation of the neck node levels for head and neck tumors: a 2013 update. DAHANCA, EORTC, HKNPCSG, NCIC CTG, NCRI, RTOG, TROG consensus guidelines. Radiother Oncol. 2014 Jan;110(1):172-81. doi: 10.1016/j.radonc.2013.10.010. Epub 2013 Oct 31. PMID 24183870